CLINICAL TRIAL: NCT06235333
Title: Exploring a Lottery-promoted Gambling Disorder Screening Day Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge Health Alliance (Other)
Collaborators: International Center for Responsible Gaming (Unknown); Hoosier Lottery, Indiana (Unknown)
Responsible Party: Principal Investigator, Debi LaPlante, Director, Division on Addiction, Cambridge Health Alliance
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 13656
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Gambling Problem
Keywords: brief screening

STUDY DESIGN:
Intervention Model Description: There are two possible conditions: (1) intervention, which consists of a branching responsible/problem gambling information and gambling screening experience and (20 control, which consists of limited responsible/problem gambling information experience.
Who Masked: Investigator
Masking Description: Through Qualtrics programming, individuals will be randomly assigned to an intervention or control group. Because this happens automatically, the investigators will not know assigned conditions until after data collection is completed. Participants will be aware of their condition because they will either participate in a screening or receive problem/responsible gambling information before completing a survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening Intervention (Experimental): Individuals will take part in a branching problem/responsible gambling information sharing experience before completing a multi-item brief gambling screen and receiving tailored feedback about their risk for gambling-related problems, and including problem/responsible gambling resources for their state of residence and national resources.
  Interventions: Behavioral: Gambling Disorder Screening Day screener
- Informational Control (Active Comparator): Individuals will take part in a limited problem/responsible gambling information sharing experience.
  Interventions: Behavioral: Gambling Disorder Screening Day information sheet

INTERVENTIONS:
Behavioral: Gambling Disorder Screening Day screener — See descriptions
  Arms: Screening Intervention
Behavioral: Gambling Disorder Screening Day information sheet — See descriptions
  Arms: Informational Control

SUMMARY:
The study is a randomized trial of gambling screening plus feedback (intervention) or gambling information (control) conditions, with data collection at baseline (T1) and a 3-month follow-up (T2). Two participant recruitment strategies (i.e., Hoosier Lottery cohort and MTurk Workers cohort) will allow the investigators to compare how recruitment source relates to post-intervention gambling behavior change intentions and assorted gambling-related behavior changes. The investigators also seek to understand how experiences with screening vary for minoritized and non-minoritized people who gamble.

DETAILED DESCRIPTION:
Gambling Disorder Screening Day (GDSD) occurs on the second Tuesday of March annually. This events is modeled after National Alcohol and Depression Screening Days, which research shows increase awareness and help-seeking for these problems. There has never been a study of the impacts of GDSD on its participants. The event is growing in popularity across Massachusetts, the U.S., and around the world, which makes its assessment imperative. Gambling operators might be able to support independent public health interventions for safer gambling due to their reach (e.g., through email marketing lists) among gamblers. Operator involvement in such efforts would help fulfill their responsibility for promoting safer gambling and help-seeking. Although limited public health expertise and opposing financial interests limit the value of operators' direct involvement in public health intervention, the value of indirect support through promoting third-party public health efforts remains an open question. Accordingly, this study considers how gambling operators might contribute to gamblers' participation in GDSD, and how it compares to another technique (e.g., MTurk) that offers high engagement.

As the event grows in popularity, it is imperative to ensure that GDSD has the intended effects, especially for high-reach supporters, such as gambling operators. This is particularly important for different types of people who might be more or less receptive to operator-promoted GDSD events. The investigators might, for example, expect to observe differences depending upon individuals' race/ethnicity status. Individuals minoritized by race/ethnicity have distinct barriers to help-seeking, including previous healthcare discrimination, lack of culturally and linguistically appropriate care, and an absence of resources and treatment opportunities designed with their unique needs and cultures in mind. Operator-promoted GDSD events, therefore, might need to be tailored to ensure reach, receptivity, and responsivity among minoritized people.

This study will provide information that can shape future gambling industry involvement in public health events, and simultaneously, complete a large (i.e., over 2,000 individuals) gambling screening. In addition, the proposed research involves a novel collaboration with an industry partner to examine a new digital protocol for gambling screening and intervention. The findings will provide new information about the efficacy of online mass screening for gambling-related problems.

Study Aims:

1. Co-develop with the Hoosier Lottery a campaign to promote a new digital protocol for gambling screening and intervention study timed to coincide with GDSD 2024 promotion;
2. Use a longitudinal sample of greater-Indiana gamblers to evaluate differences in GDSD reach (i.e., numbers of individuals screened), receptiveness (i.e., post-screening ratings of clarity, informativeness, relevance and helpfulness), and responsivity (i.e., changes in post-screening reports of gambling behavior and safer play intentions and behaviors) for lottery-recruited and platform-recruited (i.e., MTurk) screening participants randomized to intervention or control groups, using baseline and 3-month follow-up surveys and purposeful sampling; and,
3. Conduct a moderator analysis to examine whether status as a minoritized group member interacts with recruitment pathway to shape participants' responsivity to the screening/intervention protocol.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, participants must (1) be at least 18 years old, (2) have gambled at least monthly during the past 12 months, and (3) reside in Indiana, Kentucky, Michigan, Illinois, or Ohio.

Exclusion Criteria:

* Being from outside of U.S.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2024-03-12 (Estimated); Primary Completion 2024-06-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reach | Time 1 (March 12, 2024)
  At Time 1, the investigators will count the number of individuals who elect to launch the GDSD screening protocol.
Protocol Feedback. | Time 1 (March 12, 2024)
  At Time 1, the investigators will ask participants to indicate the extent to which they agree that specific parts of the GDSD protocol are (1) clear, (2) informative, (3) relevant, and (4) helpful. Participants will make ratings on a 5-point scale ranging from Strongly Disagree to Strongly Agree.
Gambling Frequency. | Time 1 (March 12, 2024) and Time 2 (June 12, 2024)
  At Time 1 and Time 2, the investigators will assess past three-months gambling behavior. The investigators will ask participants to indicate the frequency with which they engaged in six gambling activities (e.g., Lottery/Scratch Tickets; Poker, Casino Table Games; Sports; Slots/Keno; Other) in the past 3 months on a scale from Never (0) to More than Once a Week (6). For some analyses, the investigators will assign individuals a single 3-month frequency score (range 0-6) by identifying individuals' maximum frequency playing any game during the past three months.
Gambling Intentions. | Time 1 (March 12, 2024)
  At Time 1, the investigators will inquire about participants' future gambling intentions by asking them to report how much they expect they will gamble on six types of gambling games during the next three months using the same frequency scale adapted for future gambling.
Guidelines Compliance. | Time 1 (March 12, 2024) and Time 2 (June 12, 2024)
  At Time 1 and Time 2, the investigators will ask participants to report, to the best of their recollection, whether they have complied with three Lower Risk Gambling Guidelines [LRGG; 21] during the previous three months: (1) Gambled no more than 1% of household income before tax per month, (2) Gambled no more than four days per month, and (3) Avoided regularly gambling at more than two types of games.
  Participants will indicate that they have complied with a practice, have not complied, or do not know. For some analyses, the investigators will assign individuals a single compliance score (0-3) by summing the number of guidelines with which an individual complied during the past three months.
Guidelines Intentions. | Time 1 (March 12, 2024)
  At Time 1, the investigators will ask participants to report their intentions for following the three LRGG during the next three months. Participants will make ratings on a 5-point scale ranging from Extremely Unlikely to Extremely Likely.
Safer Gambling Practices. | Time 1 (March 12, 2024) and Time 2 (June 12, 2024)
  At Time 1 and Time 2, the investigators will ask participants to report, to the best of their recollection, whether they have engaged in six safer gambling practices [21] during the previous three months: (1) limit your consumption of alcohol, cannabis and other drugs while gambling; (2) limit your access to money; (3) schedule activities right after gambling sessions, which can set a limit on the amount of time you have to gamble; (4) think about how having gambling companions or gambling alone might impact you; (5) keep in mind how much money you are able to spend on entertainment when deciding how much to gamble; and, (6) plan ahead and set limits. Participants will indicate that they have engaged in a practice, have not engaged, or do not know. For some analyses, the investigators will assign individuals a single safer gambling score (0-6) by summing the number of safer gambling practices with which an individual engaged during the past three months.
Safer Gambling Intentions. | Time 1 (March 12, 2024)
  At Time 1, the investigators will ask participants to report their intentions for engaging in the six safer gambling practices during the next three months. Participants will make ratings on a 5-point scale ranging from Extremely Unlikely to Extremely Likely.
Help Seeking Behavior. | Time 1 (March 12, 2024) and Time 2 (June 12, 2024)
  At Time 1 and Time 2, the investigators will ask participants to report whether they engaged in gambling education and gambling help-seeking activities during the past three months. Participants will indicate Yes or No to whether they have engaged with (1) a gambling self-help workbook that can be completed anonymously online; (2) a gambling self-help workbook that was mailed to their home; (3) an online gambling helpchat; (4) a phone-based gambling helpline; (5) a gambling recovery podcast; (6) a gambling recovery smartphone app; (7) Gamblers Anonymous or other mutual support groups; (8) gambling "how to" books or services; or (9) professional treatment for gambling, including a more in-depth assessment of their gambling behavior. For some analyses, the investigators will assign individuals a single help seeking score (0-9) by summing the number of help-seeking activities with which an individual engaged during the past three months.
Help Seeking Intentions. | Time 1 (March 12, 2024)
  At Time 1, the investigators will ask participants to indicate their likelihood of engaging in the nine gambling education and gambling help-seeking activities during the next three months. Participants will make ratings on a 5-point scale ranging from Extremely Unlikely to Extremely Likely.
Positive Play Scale. | Time 1 (March 12, 2024) and Time 2 (June 12, 2024)
  At Time 1 and Time 2, the investigators will ask participants to complete the Positive Play Scale [22] on a 3-month timeframe. The investigators will calculate Cronbach's alpha and, if the investigators observe adequate internal consistency, the investigators will calculate its four subscale scores by summing.

CONTACTS AND LOCATIONS:
Overall Officials: Debi A. LaPlante, PhD, Principal Investigator — Cambridge Health Alliance

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share data on the Division on Addiction Transparency Project website.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Following publication of associated papers.
URL: http://www.thetransparencyproject.org